CLINICAL TRIAL: NCT00890682
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Safety and Efficacy of a Single Administration of SKY0402 for Prolonged Postoperative Analgesia in Subjects Undergoing First Metatarsal Osteotomy (Bunionectomy)
Brief Title: Study of Postoperative Analgesia in Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SKY0402C317
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Results first posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-07

CONDITIONS: Bunion; Hallux Valgus
Keywords: Bunion; Bunionectomy; Osteotomy
MeSH Terms: conditions — Bunion; Hallux Valgus | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sky0402 (Experimental): Injection of Study Drug
  Interventions: Drug: SKY0402
- Placebo (Placebo Comparator): Injection of study drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SKY0402 — Local infiltration of 8cc SKY0402
  Other Names: EXPAREL
  Arms: Sky0402
Drug: Placebo — Local infiltration of 8cc Placebo
  Other Names: saline 0.9%
  Arms: Placebo

SUMMARY:
After undergoing bunion surgery, patients are given a pain medicine injection that may last for up to several days or a placebo. Their pain and pain medicine use is then monitored.

DETAILED DESCRIPTION:
Following drug study administration, safety and efficacy assessments were conducted

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the Screening visit
* Scheduled to undergo primary unilateral first metatarsal osteotomy without hammertoe
* Female subjects must be surgically sterile or at least two years menopausal, or using an acceptable method of birth control. If of childbearing potential, have a documented negative blood or urine pregnancy test within 24 hours before surgery
* Clinical laboratory values less than or equal to twice the upper limit of normal or, if abnormal, deemed not clinically significant per the Investigator
* Ability to provide informed consent, adhere to the study visit schedule and complete all study assessments

Exclusion Criteria:

* Currently pregnant, nursing, or planning to become pregnant during the study or within one month after study drug administration
* Chronic user of analgesic medications, including taking opioid medications for more than 14 days in the last 3 months, or non-opioid pain medications more than 5 times per week
* Use of any non-steroidal anti-inflammatory drug (NSAID) including selective COX-2 inhibitor within three days of surgery
* Use of acetaminophen within 24 hours of surgery
* Use of selective serotonin reuptake inhibitors (SSRIs), gabapentin, pregabalin (Lyrica), duloxetine (Cymbalta) within three days of surgery
* Current use of systemic glucocorticosteroids or use of systemic glucocorticoids within one month of enrollment into this study
* Peripheral neuropathy including diabetic neuropathy, chemotherapy-induced neuropathy, HIV neuropathy
* History of hepatitis
* History of, suspected, or known addiction to or abuse of drugs or alcohol within the past two years
* Failure to pass urine drug screen
* Current evidence of alcohol abuse (greater than 4 units of alcohol per day: 1 unit = ½ pint of beer, 1 glass of wine or 1 oz. of spirits)
* Evidence of peripheral ischemic disease
* Type I or Type II diabetes
* Current acute or chronic medical or major psychiatric disease that, in the opinion of the Investigator, would interfere with the evaluation of study drug efficacy or safety
* Malignancy in the last 2 years, with the exception of non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix
* Administration of an investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study
* Previous participation in a SKY0402 study
* Significant medical conditions or laboratory results that, in the opinion of the Investigator, indicate an increased vulnerability to study drugs and procedures
* Current painful physical conditions or concurrent surgery other than bunionectomy that may require analgesic treatment (such as NSAID or opioid) in the postoperative period for pain that is not strictly related to the bunionectomy procedure and may confound the postoperative assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Daniels, DO, Principal Investigator — Premier Research Group Clinical Research Center
Locations (1):
- Premier Research Group, Austin, Texas, United States

REFERENCES:
- [Derived] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785
- [Derived] Golf M, Daniels SE, Onel E. A phase 3, randomized, placebo-controlled trial of DepoFoam(R) bupivacaine (extended-release bupivacaine local analgesic) in bunionectomy. Adv Ther. 2011 Sep;28(9):776-88. doi: 10.1007/s12325-011-0052-y. Epub 2011 Aug 12. PMID 21842428

RESULTS

PARTICIPANT FLOW:
Groups:
- SKY0402: Injection of 8cc SKY0402 (single dose)
- Placebo: Injection of 8cc Placebo (single dose)
Period: Overall Study
Arm/Group | SKY0402 | Placebo
Started | 97 | 96
Completed | 93 | 94
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Study Drug Injection
- Total: Total of all reporting groups
Arm/Group | Sky0402 | Placebo | Total
Number analyzed (Participants) | 97 | 96 | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 92 | 189
  >=65 years | 0 | 4 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 42.4 (12.6) | 43.2 (13.3) | 42.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 84 | 159
  Male | 22 | 12 | 34
Region of Enrollment [Number; unit: participants]
  United States | 97 | 96 | 193

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of the Numeric Rating Scale at Rest (NRS-R) Pain Intensity Scores
Description: The AUC of the NRS-R pain intensity scores from time 0 through 24 hours
  The subject was to rest for at least 5 minutes before responding to the following question, "On a scale of 0 to 10, where 0 = no pain and 10 = worst possible pain, how much pain are you having right now?"
Time Frame: 0-24 hours
Measure: Geometric Mean (Standard Error); unit: Units on a scale*hours
Groups:
- SKY0402; Placebo: Single injection of study drug
Arm/Group | SKY0402 | Placebo
Number analyzed (Participants) | 97 | 96
Units on a scale*hours | 124 (4.5) | 146 (4.6)

2. Secondary Outcome: Adverse Event Profile
Description: Participants with an Adverse Event through 72 hours or a Serious Adverse Event through 30 days
Time Frame: 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Sky0402 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/97 | 1/96
Other Adverse Events (participants affected / at risk) | 56/97 | 63/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sky0402 (N=97) | Placebo (N=96)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sky0402 (N=97) | Placebo (N=96)
Nausea (Gastrointestinal disorders) | 39 | 36
Vomiting (Gastrointestinal disorders) | 27 | 17
Dizziness (Nervous system disorders) | 11 | 25
Headache (Nervous system disorders) | 5 | 8
Somnolence (Nervous system disorders) | 5 | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No